CLINICAL TRIAL: NCT03709719
Title: A Phase II Study to Evaluate the Safety and the Efficacy of a Blinatumomab Based Consolidation and Maintenance in Patients With High-risk B-cell Precursor Acute Lymphoblastic Leukemia (BCP-ALL). GRAALL-QUEST
Brief Title: Blinatumomab in High-risk B-cell Precursor Acute Lymphoblastic Leukemia
Acronym: GRAALL-QUEST
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRAALL-QUEST
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Acute Lymphoblastic Leukemia, Adult B-Cell
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- blinatumomab (Experimental)
  Interventions: Drug: Blinatumomab Injection

INTERVENTIONS:
Drug: Blinatumomab Injection — Blinatumomab 28 μg/day : D1 to D28

SUMMARY:
The GRAALL-QUEST study is a Phase 2 study nested in the GRAALL-2014/B study (NCT02617004). The GRAALL-QUEST study evaluates the safety and the efficacy of blinatumomab-containing consolidation and maintenance therapy in patients aged 18-59 years old with high-risk B-cell precursor acute lymphoblastic leukemia (BCP-ALL) in first complete hematologic remission after one induction course of standard chemotherapy and no central nervous system (CNS) involvement at diagnosis.

High-risk patients are defined as patients with KMT2A/MLL gene rearrangement, and/or IKZF1 (Ikaros) intra-genic deletion and/or high post-induction Ig-TCR minimal residual disease (MRD) level (≥10-4). In such patients not receiving blinatumomab, 3-year hematologic relapse incidence and relapse-free survival (RFS) are estimated at 60-65% and 50% only, respectively, on the basis of historical results.

A large subset of these high-risk patients (i.e. those with post-induction MRD level ≥10-3 and/or post-consolidation MRD level ≥10-4), but not all, will also be considered as candidates for allogeneic hematopoietic stem cell transplantation (allo-HSCT) in first hematologic remission. The primary objective of the GRAALL-QUEST study is to evaluate the efficacy of adding blinatumomab to consolidation and eventually maintenance therapy in term of Relapse Free Survival (RFS). Secondary objectives are overall survival, comparison of RFS and Overall Survival (OS) in transplanted versus non-transplanted patients, MRD response and safety. Blinatumomab will be given as monthly cycles at the daily dose of 28 microg/d continuous IV infusion, together with 3 triple intra-thecal (IT) chemotherapy injections. The first cycle will start after completion of the first consolidation chemotherapy phase (corresponding to the MRD2 time-point). Patients receiving allo-HSCT will receive successive blinatumomab cycles until allo-HSCT. Patients not receiving allo-HSCT will receive a first blinatumomab cycle (cycle 1) during the second consolidation chemotherapy phase, followed by late intensification, then the third consolidation chemotherapy phase including another blinatumomab cycle (cycle 2) and maintenance chemotherapy including three additional blinatumomab cycles (cycles 3 to 5), for a total of 5 blinatumomab cycles maximum.

ELIGIBILITY:
Inclusion Criteria:

* Included in GRAALL-2014/B

  1. Whose blood and bone marrow explorations have been completed before the steroids prephase
  2. Aged 18 to 59 years old with not previously treated B-lineage-ALL (including intrathecal injections) newly diagnosed according to the WHO 2008 definition with > 20% bone marrow blasts
  3. Whose karyotype shows no t(9;22) and/or the absence in molecular biology of BCR-ABL marker
  4. With Eastern Cooperative Oncology Group (ECOG) performance status < 3
  5. With or without central nervous system (CNS) or testis involvement
  6. Without other evolving cancer (except basal cell carcinoma of the skin or "in situ" carcinoma of the cervix) or its treatment should be finished at least since 6 months
  7. Having signed a written informed consent
  8. With efficient contraception for women of childbearing age (excluding estrogens and IUS)
  9. With health insurance coverage
  10. Who have received or being receiving the steroid prephase
* With High Risk (HR) B-ALL
* ECOG ≤ 3
* In Complete Remission after one or two induction cures and having received the three blocks of consolidation N°1
* With or without allogeneic donor

Exclusion Criteria:

* With ECOG status > 3 after consolidation 1
* With abnormal laboratory values as defined below after consolidation 1

  1. Aspartate transaminase (AST) (SGOT) and/or alanine transaminase (ALT) (SGPT) ≥ 5 x ULN
  2. Total bilirubin ≥ 1.5 x ULN
  3. Creatinine ≥ 1.5 x ULN or creatinine clearance < 50 ml/min
  4. Serum amylase and lipase ≥ 1.5 x ULN
* With active uncontrolled infection, any other concurrent disease or medical condition that is deemed to interfere with the conduct of the study as judged by the investigator
* New York Heart Association (NYHA) Functional Classification 3-4 cardiac disease
* Infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus (HBsAg positive) or hepatitis C virus (anti-HCV positive)

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Estimated)
Dates: Start 2018-10-20 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival Y3 | 3 years
  Disease Free Survival at 3 years

SECONDARY OUTCOMES:
OS Y3 | 3 years
  Overall survival at 3 years
CIR Y3 | 3 years
  Cumulative incidence of relapse at 3 years
NRM | 3 years
  Non Relapse related Mortality
MRD1 | after induction or on day 1 of first consolidation
  Minimal Residual Disease
MRD2 | on day 1 of second consolidation
  Minimal Residual Disease
MRD3 | on day 1 of late intensification(or at pre Allo-SCT evaluation)
  Minimal Residual Disease
MRD4 | on day 1 of maintenance phase (or at day 100 after Allo-SCT)
  Minimal Residual Disease

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital saint Louis, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided